CLINICAL TRIAL: NCT02680431
Title: Analysis of Plasma for Diagnosis and Follow-up of Neurofibromatosis Type 1
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Juha Peltonen (Other Government)
Responsible Party: Sponsor-Investigator, Juha Peltonen, Professor, Turku University Hospital
Organization: Turku University Hospital (Other Government)
Other Study IDs: 141-1801-2015
Record Dates: First submitted 2016-01-15; First posted 2016-02-11 (Estimated); Last update posted 2016-02-11 (Estimated); Status verified 2016-02

CONDITIONS: Neurofibromatosis 1
MeSH Terms: conditions — Neurofibromatosis 1 | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Free circulating DNA extracted from blood plasma
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Neurofibromatosis 1: 10 mL venous blood sample taken from patients with type 1 neurofibromatosis
  Interventions: Other: Blood sample
- Control: 10 mL venous blood sample taken from age- and gender-matched healthy controls
  Interventions: Other: Blood sample

INTERVENTIONS:
Other: Blood sample — 10 mL venous blood sample for analysis of plasma

SUMMARY:
The purpose of this study is to find blood plasma based biomarkers of disease progression in neurofibromatosis type 1 (NF1). NF1 is associated with the development of benign cutaneous tumors as well as a variety of malignancies. Analysis of plasma DNA and chemical composition may provide tools for diagnosis and follow-up of NF1. The hypothesis of the study is that NF1-associated tumor burden and malignant transformation of tumors can be detected in plasma. To test this hypothesis, Finnish patients with NF1 are recruited and blood sample is taken. Blood plasma is separated and analyzed chemically. DNA is then also extracted and quantified.

DETAILED DESCRIPTION:
Neurofibromatosis type 1 (NF1) is a dominant hereditary multiorgan disease that causes both benign cutaneous neurofibromas and malignant tumors. Timely detection of malignant transformation in NF1 tumors is of great clinical importance. Also methods to easily monitor individual's overall tumor burden would be useful. Blood plasma is collected from NF1 patients and age- and gender-matched controls. The samples are stored at -80 C until analysis. Free circulating plasma DNA is extracted and quantified using commercial reagents. Also a previously described chemical detection method to observe overall changes in plasma composition is utilized. The analysis results are compared between NF1 patients and healthy controls, and also correlated with NF1 tumor burden and diagnosis of malignancy during five-year follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Finnish-speaking
* 18-85 years old
* For NF1 group: Diagnosis of type 1 neurofibromatosis and visit to Turku Neurofibromatosis Centre
* For control group: Suitable as an age- and gender-matched control for some of the NF1 patients

Exclusion Criteria:

* Non-Finnish-speaking
* For control group: diagnosis of neurofibromatosis type 1 or cancer

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients visiting Turku Neurofibromatosis Centre (Finland) for care of their disease. Controls are healthy volunteers from Turku area.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2016-01; Primary Completion 2020-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Ability of free circulating plasma DNA concentration and unspecific chemical detection method to predict overall tumor burden | Up to 5 years
  Tumor burden assessed by clinician on a four-level scale: 1 = 0-5 neurofibromas, 2 = 6-99 neurofibromas, 3 = 100-500 neurofibromas, 4 = over 500 neurofibromas
Ability of free circulating plasma DNA concentration and unspecific chemical detection method to predict clinical diagnosis of malignancy | Up to 5 years
  Information on clinical diagnoses is obtained from patient records

CONTACTS AND LOCATIONS:
Overall Officials: Juha Peltonen, Professor, Principal Investigator — University of Turku

IPD SHARING:
Plan to Share IPD: Undecided
Molecular biology results and relevant clinical information will be shared along publication. Some clinical information is subject to privacy issues and cannot be shared.